CLINICAL TRIAL: NCT04806555
Title: Diagnostic Value of Compression Ultrasound to Detect Acute Compartment Syndrome After Lower Limb Revascularisation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kantonsspital Aarau (Other)
Responsible Party: Principal Investigator, Andrej Isaak, Head of Vascular Surgery, Kantonsspital Aarau
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-03006
Record Dates: First submitted 2021-03-10; First posted 2021-03-19 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Compartment Syndrome of Leg
Keywords: compartment syndrome; acute limb ischemia; intra compartmental pressure; compression ultrasound; vascular surgery; limb revascularisation
MeSH Terms: conditions — Compartment Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Compression ultrasound (Experimental): All recruited patients
  Interventions: Diagnostic Test: Compression ultrasound examination

INTERVENTIONS:
Diagnostic Test: Compression ultrasound examination — After successful revascularisation for acute ischemia and clinical suspicion of acute compartment syndrome, compression ultrasound (CU) will be performed in OR followed by standard intra-compartmental measurement. Two physicians will perform two subsequent measurements of the affected limb after revascularisation. The unaffected limb will be examined once to obtain baseline elasticity ratio values. All CU examinations will be documented in PACS (picture archiving and communication system) and evaluated after ICP measurement, and if necessary, fasciotomy is performed.

SUMMARY:
Acute compartment syndrome (ACS) after revascularization for acute limb ischemia is a potentially limb-threatening condition and requires urgent fasciotomy. Compression ultrasound (CU) is an established method for measuring intravenous pressure in superficial veins and, for example, can determine central venous pressure in critically ill patients. In cadaver studies, compression ultrasound has been proven to correlate with invasive intra compartmental pressure (ICP) measurements. This study aims to determine CU's added diagnostic value compared to ICP in detecting ACS after revascularisation.

DETAILED DESCRIPTION:
Acute compartment syndrome (ACS) after revascularization for acute limb ischemia is a potentially limb-threatening condition and requires urgent fasciotomy. It occurs when the tissue pressure within a closed muscle compartment exceeds the perfusion pressure and results in muscle and nerve ischemia.

If clinically suspected, intra- compartmental pressure (ICP) is measured by inserting a needle into the area of ACS, usually the anterior tibial muscle compartment, while an attached pressure monitor records the pressure. This invasive diagnostic method is widely used as a standard with a sensitivity of 94% and specificity of 98%.

Compression ultrasound (CU) is an established method for measuring intravenous pressure in superficial veins and, for example, can determine central venous pressure in critically ill patients. An ultrasound translucent probe measures the pressure applied on the skin surface with the ultrasound transducer. In cadaver studies, compression ultrasound has been proven to correlate with invasive ICP measurements. The elasticity ratio (ER, compartment diameter with and without external pressure) validated in a recently published animal model has a sensitivity of 94.4% and a specificity of 88.9% to diagnose a compartment syndrome properly. The first results in six trauma patients showed that the ER less than 10,5% of the anterior tibial compartment had a sensitivity of 95,8% and a specificity of 87,5% to an appropriate diagnosis of ACS. Thus, this non-invasive, low-cost, and secure diagnostic technique has not been validated in patients with ACS after revascularisation for acute lower limb ischemia yet has the potential to discriminate clinically suspected ACS sensitively.

This study aims to determine CU's added diagnostic value compared to ICP in detecting ACS after revascularisation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of acute compartment syndrome after revascularisation of lower limb

Exclusion Criteria:

* Not fulfilling any of the inclusion criteria
* Patients refusing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Elasticity ratio (ER) | baseline
  Sensitivity and specificity of elasticity ratio measured by compression ultrasound for detecting high intra compartmental pressure

SECONDARY OUTCOMES:
Inter- and intra-rater reliability | baseline
  Inter- and intra-rater reliability of compression ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Isaak, Dr.med., Principal Investigator — Kantonsspital Aarau
Locations (1):
- Kantonsspital Aarau, Aarau, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thalhammer C, Aschwanden M, Odermatt A, Baumann UA, Imfeld S, Bilecen D, Marsch SC, Jaeger KA. Noninvasive central venous pressure measurement by controlled compression sonography at the forearm. J Am Coll Cardiol. 2007 Oct 16;50(16):1584-9. doi: 10.1016/j.jacc.2007.07.022. Epub 2007 Oct 1. PMID 17936158
- [Background] Thalhammer C, Segerer S, Augustoni M, Jacomella V, Clemens RK, Wuthrich RP, Amann-Vesti BR, Husmann M. Acute effects of haemodialysis on central venous and arterial pressure characteristics. Nephrology (Carlton). 2015 Feb;20(2):91-5. doi: 10.1111/nep.12356. PMID 25346188
- [Background] Bloch A, Tomaschett C, Jakob SM, Schwinghammer A, Schmid T. Compression sonography for non-invasive measurement of lower leg compartment pressure in an animal model. Injury. 2018 Mar;49(3):532-537. doi: 10.1016/j.injury.2017.11.036. Epub 2017 Nov 27. PMID 29195681
- [Background] Sellei RM, Wollnitz J, Reinhardt N, de la Fuente M, Radermacher K, Weber C, Kobbe P, Hildebrand F. Non-invasive measurement of muscle compartment elasticity in lower limbs to determine acute compartment syndrome: Clinical results with pressure related ultrasound. Injury. 2020 Feb;51(2):301-306. doi: 10.1016/j.injury.2019.11.027. Epub 2019 Nov 21. PMID 31784057